CLINICAL TRIAL: NCT06406257
Title: Effect of Intraoperative Temperature Management on Postoperative Delirium in Elderly Patients Undergoing Hip Surgery
Brief Title: Temperature Management on Postoperative Delirium
Acronym: POD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wang Hongjian (Other)
Collaborators: The Second Hospital of Anhui Medical University (Other)
Responsible Party: Sponsor-Investigator, Wang Hongjian, Attending doctor, Second People's Hospital of Hefei City
Organization: Second People's Hospital of Hefei City (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2024-keyan-045
Record Dates: First submitted 2024-05-02; First posted 2024-05-09 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Emergence Delirium
Keywords: Postoperative Delirium; Body Temperature; Hyperthermia; Hypothermia
MeSH Terms: conditions — Emergence Delirium; Hyperthermia; Hypothermia

STUDY DESIGN:
Intervention Model Description: Enrolled participants were randomly assigned to a control group (Group C) or a body temperature protection group (Group W) in a 1:1 ratio.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group C (No Intervention): Patients in Group C will be covered with a bedsheet intraoperatively without active warming methods employed.
- Group W (Experimental): Patients in Group W will have a 37°C forced-air warming blanket initiated upon entering the operating room to maintain their body temperature between 36-37 degrees Celsius.
  Interventions: Device: 3M™ Bair Hugger™ Warming Unit

INTERVENTIONS:
Device: 3M™ Bair Hugger™ Warming Unit — Utilizing the 3M Temperature Management Unit to ensure intraoperative body temperature of elderly hip surgery patients remains consistent with their preoperative baseline, while patients in Group C receive no intervention.
  Arms: Group W

SUMMARY:
Presently, the effects of perioperative temperature management on postoperative delirium remain ambiguous. This study endeavors to explore the influence of intraoperative temperature variations in elderly hip fracture patients on postoperative delirium.

DETAILED DESCRIPTION:
At present, the pathophysiological mechanisms contributing to postoperative delirium in elderly hip fracture patients remain elusive, with predominant research concentrating on neural inflammation, neurotransmitter dysregulation, and metabolic irregularities. The influence of perioperative temperature management on postoperative delirium remains uncertain and may correlate with surgical modality and intraoperative temperature modulation. Hence, this study endeavors to juxtapose intraoperative temperature variations among elderly hip fracture patients, probing their ramifications on postoperative delirium.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* Classified as American Society of Anesthesiologists I-III
* Hip surgery patients who agreed to the study

Exclusion Criteria:

* Non-consent to participate
* Diagnosed neurological or psychiatric disorders including schizophrenia, epilepsy, Parkinson's disease, or myasthenia gravis
* Coma, dementia, or language impairment affecting communication and assessment
* History of neurosurgery
* Use of antipsychotic medication preoperatively
* Body temperature exceeding 38°C within 24 hours before surgery.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-05-20 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | Within 3 days after surgery
  Confusion Assessment Method (CAM) was recorded before surgery, 10 min after admission to PACU, before exiting the post-anesthesia care unit (PACU), and 1, 2, and 3 days after surgery. POD was diagnosed if the patient had at least one episode of delirium at these time points after surgery.
  The CAM diagnostic algorithm is based on four cardinal features of delirium: 1) acute onset and fluctuating course, 2) inattention, 3) disorganized thinking, and 4) altered level of consciousness. A diagnosis of delirium according to the CAM requires the presence of features 1, 2, and either 3 or 4.

SECONDARY OUTCOMES:
Incidence of intraoperative hypothermia | During operation
  Perioperative hypothermia was defined as a drop in core temperature below 36 ℃. Intraoperative tympanic membrane temperature was measured to record the incidence and duration of hypothermia.
Pleiotropic cytokine in the patient's serum | Serum interleukin-6 (IL-6) levels before surgery and at 1, 2, and 3 days after surgery.
  Clinical trials and meta-analyses have identified the association between POD and increased perioperative levels of Interleukin-6 (IL-6), a pleiotropic cytokine that is both necessary and sufficient for postoperative memory decline in a preclinical model of POD.

CONTACTS AND LOCATIONS:
Overall Officials: Xianwen Hu, PhD, Study Chair — The Second Hospital of Anhui Medical University

IPD SHARING:
Plan to Share IPD: No
Currently, it remains unclear how IPD sharing will be conducted.